CLINICAL TRIAL: NCT05569226
Title: OKKO Health Hyperacuity, Contrast and Colour Game Validation in Age-related Macular Degeneration
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: OKKO Health (Industry)
Responsible Party: Sponsor
Other Study IDs: OKHR-07
Record Dates: First submitted 2022-10-03; First posted 2022-10-06 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Smartphone apps have the potential to measure standard metrics of visual function. In addition, new tests may serve as digital biomarkers to detect early progression of disease, assess risk of developing disease or expand the patient's clinical picture. Smartphones are inherently advantageous to reduce the reliance on specialist bulky and costly equipment that currently only exists in specialist clinics. While there are some smartphone apps available for vision monitoring, very few have any clinical evidence to support reliability, validity and diagnostic accuracy.

The OKKO Health app (www.okkohealth.com) is a smartphone app available on Apple iOS and Android platforms, consisting of short games with applied vision science technology to measure visual function in an engaging way. The app has one game per function, each on average 1-2 minutes. There are 4 game modes available testing visual acuity, contrast sensitivity, colour sensitivity and hyperacuity. This study will aim to validate these measures of visual function against gold standard clinical tests.

ELIGIBILITY:
Inclusion Criteria:

* Participants with AMD in at least one eye
* Willing to travel to the clinic in Exmouth/Bristol
* Able to hold and use a smartphone

Exclusion Criteria:

* Significant ocular pathology other than AMD
* Unable to provide written informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People with dry or wet age-related macular degeneration.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | Day 1
  Visual acuity collected in the OKKO Health app and via ETDRS chart
Contrast sensitivity | Day 1
  Contrast sensitivity collected in the OKKO Health app and via Pelli Robson chart.
Colour sensitivity | Day 1
  Colour sensitivity collected in the OKKO Health app and via City University colour test/Mollon-Reffin colour vision test.

SECONDARY OUTCOMES:
Visual distortion | Day 1
  Visual distortion assessed using the OKKO Health app and Amsler chart.
Optical coherence tomography (OCT) | Day 1
  Scans obtained from OCT.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Kawadler, PhD, Principal Investigator — OKKO Health
Locations (1):
- Bristol, Bristol, United Kingdom